CLINICAL TRIAL: NCT07063485
Title: A Comprehensive Approach Integrating Resilience Theory and Satir Model Nursing Skills Training for Adolescent Depression: A Randomized Controlled Trial
Brief Title: Resilience and Satir Model Training for Adolescent Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Kenan Ren, Principal investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021S00495
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Adolescent Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Resilience Theory and Satir Model Nursing Skills Training Group (Experimental): Participants in this group received routine nursing care plus a specialized intervention combining resilience theory and Satir model nursing skills training. The intervention was delivered in a hospital setting and included 15 group activity sessions (2 hours each). Activities were conducted in a workshop format with fixed themes such as "I am a unique existence," "resilient beliefs," and "identifying inner sources of resilience." The sessions incorporated experiential interactive learning, progressive muscle relaxation training, and guided imagery. After each activity, participants completed tasks and shared experiences. Post-discharge follow-up was conducted to monitor progress.
  Interventions: Behavioral: Resilience Theory and Satir Model Nursing Skills Training
- Active Comparator: Routine Intervention Group (Active Comparator): Participants in this group received routine nursing intervention. This included observation of the illness condition, guidance on daily life and diet, psychological care, and health education about the disease for both patients and their families. They were also guided on emotion regulation, sleep, and medication routines, with encouragement for regular outpatient follow-ups.
  Interventions: Behavioral: Routine Nursing Intervention

INTERVENTIONS:
Behavioral: Resilience Theory and Satir Model Nursing Skills Training — A structured psychological and nursing intervention program based on resilience theory and the Satir model. It consists of 15 two-hour group sessions during hospitalization, focusing on enhancing resilience, communication, and self-efficacy through themed activities, interactive learning, relaxation techniques, and guided training. The intervention is led by psychologists and psychiatric nurses and includes post-discharge follow-up.
  Arms: Experimental: Resilience Theory and Satir Model Nursing Skills Training Group
Behavioral: Routine Nursing Intervention — Standard nursing care for patients with depression, including illness monitoring, daily life guidance, psychological support, and health education on disease management, emotion regulation, and medication.
  Arms: Active Comparator: Routine Intervention Group

SUMMARY:
This randomized controlled trial aims to assess the effectiveness of an intervention combining resilience theory with Satir model nursing skills training compared to routine nursing care for adolescents with depression. The study evaluates changes in depressive symptoms, psychological resilience, self-esteem, coping styles, and medication adherence.

DETAILED DESCRIPTION:
Adolescent depression is a growing mental health concern with significant impacts on academic and social functions. While psychological interventions are crucial, conventional methods may have limitations. This study introduces and evaluates a novel intervention that integrates resilience theory, focusing on patients' strengths and potential, with the Satir model, which addresses psychological issues from individual, family, and social systems. The study randomized 182 adolescents with depression into two groups: a research group receiving the integrated intervention and a control group receiving routine nursing care. The primary objective is to determine if the comprehensive intervention is more effective in alleviating depressive symptoms and improving psychological well-being, including resilience, self-esteem, and coping mechanisms. The findings aim to provide evidence for a new, effective therapeutic strategy for this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis aligning with the ICD-10 criteria for depressive episodes.
* First onset with a course between 4 weeks and 12 months.
* Age between 13 and 18 years.
* Normal communication ability.
* No antidepressant use in the four weeks preceding admission, and no prior psychological treatment.
* HAMD-24 score exceeding 20 points.
* Informed consents from family members or guardians.

Exclusion Criteria:

* Participants withdrawing prematurely.
* Presence of organic lesions.
* Antidepressant or psychological treatment before enrollment.
* Allergic constitution.
* Depression induced by physical illness.
* Suicide ideation score ≥4 points in MADRS with suicidal tendency.
* Diagnosis of bipolar affective disorder.
* Coexistence of other mental illnesses.
* Neurological diseases or substance dependence/abuse.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 182 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Depressive Symptoms as measured by the 17-item Hamilton Depression Scale (HAMD-17) | Baseline (at admission) and 3 Months Post-intervention
  The HAMD-17 is a clinician-rated scale with 17 items scored on a 0-4 or 0-2 point scale. A higher total score indicates more severe depressive symptoms.
Change in Depressive Symptoms as measured by the Montgomery-Åsberg Depression Rating Scale (MADRS) | Baseline (at admission) and 3 Months Post-intervention
  The MADRS is a 10-item clinician-rated scale, with each item scored from 0-6. The total score ranges from 0-60, with higher scores indicating more severe depression.
Change in Depressive Symptoms as measured by the Beck Depression Inventory (BDI) | Baseline (at admission) and 3 Months Post-intervention
  The BDI is a 13-item self-report questionnaire where items are scored from 0-3. Higher total scores indicate more severe depression.

SECONDARY OUTCOMES:
Change in Psychological Resilience as measured by the Resilience Scale for Chinese Adolescents (RSCA) | Baseline (at admission) and 3 Months Post-intervention
  The RSCA is a 27-item scale assessing five dimensions: interpersonal assistance, family support, positive cognition, emotional control, and goal focus. The total score ranges from 27 to 135. Higher scores indicate higher levels of psychological resilience.
Change in Self-Esteem Level as measured by the Feelings of Inferiority Scale (FIS) | Baseline (at admission) and 3 Months Post-intervention
  The FIS is a 36-item scale assessing dimensions of self-esteem, social confidence, learning ability, appearance, and experience, scored from 0-6. A higher score indicates stronger self-esteem.
Change in Coping Styles as measured by the Simplified Coping Style Questionnaire (SCSQ) | Baseline (at admission) and 3 Months Post-intervention
  The SCSQ is a 20-item questionnaire measuring positive coping (12 items) and negative coping (8 items). Scores range from 0-3. Higher scores on each subscale indicate a greater inclination toward that coping style.
Change in Medication Compliance as measured by the Medication Adherence Rating Scale (MARS) | Baseline (at admission) and 3 Months Post-intervention
  The MARS is a 10-item scale assessing medication compliance behaviors and attitudes. The total score ranges from 0 to 10. A higher score indicates better medication compliance.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China